CLINICAL TRIAL: NCT04119180
Title: Sedation Versus Protective Stabilization for Dental Treatment of Children With Caries and Negative Behavior at the Dentist: a Non-randomized Clinical Trial
Brief Title: Sedation Versus Protective Stabilization for Pediatric Dental Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: University of Sao Paulo (Other); King's College London (Other)
Responsible Party: Principal Investigator, Luciane Ribeiro de Rezende Sucasas da Costa, Professor, Universidade Federal de Goias
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI03925-2019; 424339/2018-8 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2019-10-01; First posted 2019-10-08 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Child Behavior; Dental Caries in Children
Keywords: Dental Anxiety; Dental Caries; Conscious Sedation; Physical Restraint; Cost-Efficacy Analysis
MeSH Terms: conditions — Child Behavior; Dental Caries | interventions — Ketamine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation (Experimental): The child receives sedatives approved for use in an outpatient setting, directed by a doctor, to accomplish the dental treatment.
  Interventions: Drug: Ketamine 50 MG/ML; Drug: Midazolam Hcl 2Mg/Ml Syrup
- Control (Other): The child does not receive sedatives. As s/he exhibits negative behavior for the dental procedure, s/he will be restrained by a family member and dental team.
  Interventions: Procedure: Protective stabilization

INTERVENTIONS:
Drug: Ketamine 50 MG/ML — Ketamine injectable solution in a concentration of 50.0 mg/mL via oral route; dose of 4.0 mg/kg maximum 100.0 mg
  Other Names: Ketamin S, Cristalia, São Paulo, Brazil
  Arms: Sedation
Drug: Midazolam Hcl 2Mg/Ml Syrup — Midazolam oral solution in a concentration of 2.0 mg/mL via oral route; dose of 0.5 mg/kg, maximum 5.0 mg when associated with ketamine;
  Other Names: Dormire oral solution, Cristalia, Sao Paulo, Brazil
  Arms: Sedation
Procedure: Protective stabilization — The legal guardian or accompanying person appointed by the legal guardian should sit in the dental chair with the child and contain leg and arm movements. A dental assistant keeps the child's head contained during care.
  Arms: Control

SUMMARY:
There is a lack of evidence on the effectiveness of moderate sedation in pediatric dentistry, compared to protective stabilization, which remains routinely used in the Brazilian context despite moral questions. The objective of this prospective nonrandomized clinical trial is to evaluate the effectiveness of the use of moderate sedation, compared to the protective stabilization, in the dental care of children with fear / anxiety and / or dental behavior problem, and associated factors. The study will be carried out in outpatient clinics of the Dental Schools of the Federal University of Goiás (UFG) and University of São Paulo (USP), with the support of professors from King's College London through the partnership CEDACORE - Children Experiencing Dental Anxiety: Collaboration on Research and Education. Participants will be 152 children under 7 years of age with dental caries, who need specialized dental treatment due to a history of non-cooperation with dental care. The interventions to be compared are moderate sedation with oral administration of ketamine and midazolam (UFG) and protective stabilization (USP). The primary endpoint 'behavior / anxiety of the child during treatment will be assessed using the Ohio State University Behavioral Rating Scale. The secondary outcomes are: dental behavioral and anxiety evolution of the child, child' pain during procedure, impact on the quality of life related to oral health, parents and dentists' satisfaction and stress, adverse events for sedated participants, longevity of composite and glass ionomer cement restorations, chronotype and physiological stress of these children. A cost-efficacy analysis will be produced at the end of the study from the perspective of the Sistema Único de Saúde. Additionally, at the end of 36 months, the investigators expect to contribute to the identification of psychosocial aspects related to dental behavior problems in children in early childhood. It is important to highlight the perspective of technological innovation, with the creation of a digital platform that will allow the registration of data related to the dental care of children worldwide and favor analyzes in the methodology of data science.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting cavities that need dental restoration
* ASA I (healthy) or II (mild and controlled systemic disease - persistent asthma, for example) children (ASA, 2015)
* Medical history without neurological or cognitive impairment
* Children who do not use medicines that may impair cognitive functions
* Children at low risk for airway obstruction (Mallampati less than 2 and / or tonsil hypertrophy occupying less than 50% of the oropharynx) (Mallampati et al., 1985)

Exclusion Criteria:

* Children with positive or definitely positive behavior (Frankl et al. 1962) in the dental examination session
* Non-attendance at the first intervention appointment after three scheduling attempts
* Chronic use of systemic corticosteroids

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Child behavior during the dental treatment | Participants will be followed for the duration of the dental session, an expected average of 40 minutes
  Children's behavior assessed by OSUBRS (Ohio State University Behavioral Rating Scale) in digital videos recorded during the administration. Scores: 1 - quiet, 2 - cry with movement, 3 - movement without cry; 4 - struggling. The higher the percentage of time of care in which the child behaves quietly, the better their behavior. Measurements for each group will be synthesized as mean (or median) and standard deviation (or interquartile range).

SECONDARY OUTCOMES:
Progression of child behavior throughout the follow-up | Baseline (dental examination) plus follow-up sessions at 4, 8, and 12 months post-treatment
  A 10-centimeter Visual Analogue Scale (VAS) is used by one of the trained/calibrated dentists to measure the child behavior during the dental session (Hosey and Blinkhorn, 2005). The VAS anchors are "negative behavior" (left) and "positive behavior" (right). At the end of the session, raters mark a point on the 10 cm line to correspond to the perceived level of behavior; this is then measured using a ruler to give a score to the nearest millimeter which can vary from 0 to 100). The higher the VAS score, the better the child's behavior assessed by the dentist
Progression of child dental anxiety throughout the follow-up | Baseline (dental examination) plus follow-up sessions at 4, 8, and 12 months post-treatment
  Facial Image Scale (Buchanan and Niven, 2002), a row of five faces ranging from "very happy" to "very sad," and numbered from 1 (very happy, most positive response) to 5 (very sad, the most negative).
Impact on oral health-related quality of life and changes after treatment | Baseline (dental examination) plus follow-up sessions at 4, 8, and 12 months post-treatment
  The B-ECOHIS is a measure of oral health-related quality of life (OHRQoL) validated in Brazil by Scarpelli et al. (2008) to assess the impact of oral health problems and related treatment on the quality of life of children aged zero to five years and their families. "The ECOHIS consists of 13 questions divided into two main parts: child impact section (part one) and family impact section (part two). The child impact section comprises of four subscales: child symptom, child function, child psychology and child self-image/social interaction. The family impact section contains two subscales: parental distress and family function. The questionnaire is scored using a simple five-point Likert scale with responses ranging from "never" to "very often" (equivalent to a score of 0 and 4, respectively). A total score ranging from zero to 52 is calculated as a simple sum of the responses with higher scores denoting a greater oral health impact and/or poorer OHRQoL." (Martins-Junior et a. 2012).
Parental satisfaction with the intervention | At the end of each session from dental examination through the end of the dental treatment, an average of 2 months
  A 10-centimeter Visual Analogue Scale (VAS) is used by the accompanying adult to measure her/his satisfaction with the child's dental session. The VAS anchors are "no satisfaction" (left) and "extreme satisfaction" (right). At the end of the session, raters mark a point on the 10 cm line to correspond to their level of satisfaction; this is then measured using a ruler to give a score to the nearest millimeter, which can vary from 0 to 100. The higher the VAS score, the greater the respondent satisfaction
Parental stress (anxiety) with the intervention | At the end of each session from dental examination through the end of the dental treatment, an average of 2 months
  A 10-centimeter Visual Analogue Scale (VAS) is used by the accompanying adult to measure her/his perceived stress (anxiety) with the child's dental session. The VAS anchors are "relaxed" (left) and "too nervous" (right). At the end of the session, raters mark a point on the 10 cm line to correspond to their level of stress (anxiety); this is then measured using a ruler to give a score to the nearest millimeter, which can vary from 0 to 100. The higher the VAS score, the greater the respondent stress
Dentist's satisfaction with the intervention | At the end of each session from dental examination through the end of the dental treatment, an average of 2 months
  A 10-centimeter Visual Analogue Scale (VAS) is used by the dentist in charge to measure her/his satisfaction with the child's dental session. The VAS anchors are "no satisfaction" (left) and "extreme satisfaction" (right). At the end of the session, raters mark a point on the 10 cm line to correspond to their level of satisfaction; this is then measured using a ruler to give a score to the nearest millimeter, which can vary from 0 to 100. The higher the VAS score, the greater the respondent satisfaction
Dentist's stress (anxiety) with the intervention | At the end of each session from dental examination through the end of the dental treatment, an average of 2 months
  A 10-centimeter Visual Analogue Scale (VAS) is used by the dentist in charge to measure her/his perceived stress (anxiety) with the child's dental session. The VAS anchors are "relaxed" (left) and "too nervous" (right). At the end of the session, raters mark a point on the 10 cm line to correspond to their level of stress (anxiety); this is then measured using a ruler to give a score to the nearest millimeter, which can vary from 0 to 100. The higher the VAS score, the greater the respondent stress
Child pain reported by the parent | At the end of each session from dental examination through the end of the dental treatment, an average of 2 months
  A 10-centimeter Visual Analogue Scale (VAS) is used by the accompanying child to measure her/his perceived pain in the child undergoing dental treatment. The VAS anchors are "no pain" (left) and "too much pain" (right). At the end of the session, raters mark a point on the 10 cm line to correspond to the perceived level of child's pain; this is then measured using a ruler to give a score to the nearest millimeter, which can vary from 0 to 100. The higher the VAS score, the greater the child's pain according to the parent
Child pain reported by the dentist | At the end of each session from dental examination through the end of the dental treatment, an average of 2 months
  A 10-centimeter Visual Analogue Scale (VAS) is used by the dentist in charge to measure her/his perceived pain in the child undergoing dental treatment. The VAS anchors are "no pain" (left) and "too much pain" (right). At the end of the session, raters mark a point on the 10 cm line to correspond to the perceived level of child's pain; this is then measured using a ruler to give a score to the nearest millimeter, which can vary from 0 to 100. The higher the VAS score, the greater the child's pain according to the dentist
Child pain/distress during the dental restoration session | Duration of the dental session, an expected average of 40 minutes
  FLACC Pain Assessment Tool (Faces, Legs, Activity, Cry and Consolability) scored by trained and calibrated observers after watching the videos of the dental treatment. The FLACC is a measurement used to assess pain for children between the ages of 2 months and 7 years. The scale is scored in a range of 0-10 with 0 representing no pain and 10, too much pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2: face, legs, activity, cry and consolability (Merkel et al., 1997).
Adverse events during the dental procedure | Participants will be followed for the duration of the dental session, an expected average of 40 minutes. Sedated patients will also be followed in the recovery room, an expected average of 60 minutes
  Occurrence of adverse events assessed by the Tracking and Reporting Outcomes of Procedural Sedation (TROOPS) (Roback et al. 2018) in the Moderate Sedation Group, or occurrence of bruises or inconsolability in the protective stabilization group
Number of teeth restored | End of each session of dental treatment, an average of 2 months
  Restored teeth count at the end of each session
Longevity of composite resin and glass ionomer cement restorations | At a time point of 5 minutes (average) after the end of the dental procedure, and in the follow-up sessions (4, 8 and 12 months)
  Trained and calibrated observers will follow the criteria for assessing occlusal (Frencken and Holmgren 2001) or occlusal-proximal (Roeleveld et al. 2006) restorations to categorize each restoration as successful or failed
Children's stress according to salivary cortisol | Change from baseline in the salivary cortisol at an expected average of 40 minutes
  Occurrence of stress during dental procedure, assessed by salivary cortisol in children; the ELISA test will determine changes in cortisol level during dental treatment
Cost analysis | An expected average of 15 months
  Cost-efficacy of different sedation protocols according to the methodology of health technologies assessment; the cost of each intervention will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Luciane RS Costa, PhD, Principal Investigator — Universidade Federal de Goias; Daniela P Raggio, PhD, Study Director — University of Sao Paulo; Patricia C Faria, PhD, Principal Investigator — Universidade Federal de Goias
Locations (2):
- Brazil (2):
  - Dental School - UFG, Goiânia, Goiás
  - Dental School - FOUSP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: 2023 to 2024
Access Criteria: According to the digital platform rules.

REFERENCES:
- [Derived] da Silva GS, Anabuki AA, Viana KA, Correa-Faria P, Moterane MM, Tedesco TK, Costa PS, Hosey MT, Raggio DP, Costa LR; CEDACORE Collaborative Group. Sedation versus protective stabilization for dental treatment of children with caries and challenging behavior at the dentist (CHOOSE): a study protocol for a non-randomized clinical trial. BMC Oral Health. 2021 May 12;21(1):256. doi: 10.1186/s12903-021-01594-0. PMID 33980232
- Available data/document: Study Protocol — https://bmcoralhealth.biomedcentral.com/articles/10.1186/s12903-021-01594-0